CLINICAL TRIAL: NCT05067998
Title: The Benefits of Natural Medicine, Vitamin IV Therapy and Supplements: Maintaining Good Health Through Nature
Status: Recruiting | Type: Observational
Sponsor: Faith A. Richardson (Other)
Responsible Party: Sponsor-Investigator, Faith A. Richardson, Psychotherapist/Licensed Holistic Health Practitioner, The Essence of Integrative Health and Medicine Practice
Organization: The Essence of Integrative Health and Medicine Practice (Other)
Other Study IDs: NatIVSup
Record Dates: First submitted 2021-09-19; First posted 2021-10-05 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Anxiety Disorders and Symptoms; Fibromyalgia; Arthritis; Chronic Pain; Hypertension,Essential
MeSH Terms: conditions — Anxiety Disorders; Fibromyalgia; Arthritis; Chronic Pain; Essential Hypertension | interventions — Phytotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Week
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (4):
- IV Vitamin Therapy Treatments: IV vitamin infusion therapy involves inserting an IV line into a vein in your arm to administer a high concentration of liquid vitamins, antioxidants, amino acids, and minerals into your bloodstream. The therapy may be for only one vitamin or a cocktail of nutrients.
  Interventions: Dietary Supplement: IV Vitamin Infused Therapy Treatment
- Herbal Medicine, Tincture (Liquid Vitamins): Tinctures are concentrated herbal extracts made by soaking the bark, berries, leaves (dried or fresh), or roots from one or more plants in alcohol or vinegar. The alcohol or vinegar pulls out the active ingredients in the plant parts, concentrating them as a liquid. Examples of common herbal health products and supplements include black cohosh, echinacea, garlic, ginkgo, saw palmetto, and St. John's wort. Herbal Medicine is type of medicine that uses roots, stems, leaves, flowers, or seeds of plants to improve health, prevent disease, and treat illness.
  Interventions: Dietary Supplement: IV Vitamin Infused Therapy Treatment
- Supplements: Dietary supplements are substances you might use to add nutrients to your diet or to lower your risk of health problems such as osteoporosis or arthritis. Dietary supplements come in the form of pills, capsules, powders, gel capsules and tablets, extracts, or liquids. Dietary supplements come in a variety of forms, including tablets, capsules, gummies, and powders, as well as drinks and energy bars. Popular supplements include vitamins D and B12; minerals like calcium and iron; herbs such as echinacea and garlic; and products like glucosamine, probiotics, and fish oils.
  Interventions: Drug: Herbal medicine
- Vitamins (Orally): Vitamins are substances that our bodies need to develop and function normally. They include vitamins A, C, D, E, and K, choline, and the B vitamins (thiamin, riboflavin, niacin, pantothenic acid, biotin, vitamin B6, vitamin B12, and folate/folic acid). Vitamins are essential nutrients that enable your body to work properly and to stay healthy. Most vitamins can be found in the food that we eat or from vitamin supplements.
  Interventions: Drug: Herbal medicine

INTERVENTIONS:
Dietary Supplement: IV Vitamin Infused Therapy Treatment — Vitamin B, C, D, E, K, liquid vitamins, antioxidants, amino acids, and minerals
  Groups: Herbal Medicine, Tincture (Liquid Vitamins); IV Vitamin Therapy Treatments
Drug: Herbal medicine — Herbal medicine is the use of plants to treat disease and enhance general health and wellbeing. Examples of common herbal health products and supplements include black cohosh, echinacea, garlic, ginkgo, saw palmetto, and St. John's wort just to name a few.
  Groups: Supplements; Vitamins (Orally)

SUMMARY:
Herbal Medicine is known as the medicinal use of herbal substances as a means of treating different conditions in the human body to ensure that the body remains in optimal health and wellness. These substances are known to contain very active ingredients in it and as such is also a very potent means of managing diseases and ailments in the body.

Herbal medicine has always been a standby source of getting relief from various conditions over centuries, however, it can be categorically said that the mode of usage of these herbal substances has changed over time. Traditional healers help individuals to make meaning out of the natural herbs seen around that can be useful to one's health.

Herbal medicine is the use of plants to treat disease and enhance general health and wellbeing. Herbs can interact with other pharmaceutical medications and should be taken with care. Always seek a regular medical doctor (GP) about any health concerns and tell them about any herbal medicines you are taking or thinking of taking. Never stop taking prescribed medications in favor of herbs without first discussing it with your GP.

DETAILED DESCRIPTION:
The major use of herbal medicines is for health promotion and therapy for chronic, as opposed to life-threatening, conditions. However, usage of traditional remedies increases when conventional medicine is ineffective in the treatment of disease, such as in advanced cancer and in the face of new infectious diseases.

Some popular options include vitamin C, B12, and, increasingly, vitamin D, while also offering vitamin D3 drips. Vitamin D, sometimes called the "sunshine vitamin" because it can be obtained through sun exposure, helps the body absorb calcium, according to the National Institutes of Health. Some people may be turning to drips of the vitamin because they aren't getting their share of sunshine this time of year and because they want to maintain a strong and healthy immune system.

Vitamin D3 is the version to go for since the body absorbs it better than vitamin D2, Taub-Dix says. But she advises against getting your vitamin D from an IV and instead shop for an oral supplement, since it's readily available on pharmacy and grocery store shelves and is easy to take by mouth. It's safe to take at dosages of up to 4,000 international units (IU). IV therapy has recently enjoyed a spike in popularity in people who rely on it as a sure-fire way to obtain all the health benefits and vitamins necessary to help them combat ailments as well as to feel their best as they cope with the pandemic.

There are several types of intravenous vitamin therapies and vitamin injections to choose from. The ones containing a large assortment of vitamins necessary to combat the flu are in highest demand. These are the ones containing Vitamin C, D, Zinc, and Vitamin B12 - all of which are vitamins known to play an essential role in assisting the body in its production of red blood cells and common immune system boosters.

"The benefit of IV therapy is that by intravenously or intramuscularly administering vitamins, you are able to absorb 100 percent of what is being put in versus supplements which must be broken down. The therapy itself only takes about 30 minutes to an hour and is monitored. Once the infusion is finished, the IV is removed and the person who received the treatment is free to go home without restrictions.

Intravenous vitamin therapy has proven helpful in the treatment of several different conditions that affect not only the immune system but other parts of the body as well. Some of the ailments of this type of therapy can help with constant fatigue, headaches, "brain fog" dry or tired looking skin, dehydration or frequent illness.

For years, people have turned to Vitamin C pills or multivitamins to help boost their immune systems. But with IV therapy, the options are endless.

If we are looking to strengthen our body and give our immune system a boost, intravenous IV therapy is the best option to do so, quickly and effectively. The body needs many different types of vitamins and nutrients to maintain normal function throughout day to day life. However, the body cannot create these vitamins on its own. Most vitamins and nutrients come from external sources, mostly from what we eat and drink. However, as efficient as the metabolic process is, the body does not absorb all the nutrients. IV therapy circumvents this problem and ensures 100% absorption because the nutrients are delivered directly into the bloodstream.

The effectiveness of IV drip therapy is especially valuable during illness, when the body's demand for nutrients is greater than usual. Supplements are invaluable to the healing process and helping the body recover more quickly.

Drip Hydration offers many IV drip therapy options to quickly and effectively improve the symptoms of a wide variety of conditions. There will also custom-blend formulas upon request. Each of our treatments contain a unique combination of ingredients. Intravenous administration of nutrients can achieve serum concentrations not obtainable with oral, or even intramuscular (IM), administration. For example, as the oral dose of vitamin C is increased progressively, the serum concentration of ascorbate tends to approach an upper limit, as a result of both saturation of gastrointestinal absorption and a sharp increase in renal clearance of the vitamin. (3) When the daily intake of vitamin C is increased 12-fold, from 200 mg/day to 2,500 mg/day, the plasma concentration increases by only 25 percent, from 1.2 to 1.5 mg/dL. The highest serum vitamin C level reported after oral administration of pharmacological doses of the vitamin is 9.3 mg/dL. In contrast, IV administration of 50 g/day of vitamin C resulted in a mean peak plasma level of 80 mg/dL. (4) Similarly, oral supplementation with magnesium results in little or no change in serum magnesium concentrations, whereas IV administration can double or triple the serum levels, (5,6) at least for a short period of time.

Various nutrients have been shown to exert pharmacological effects, which are in many cases dependent on the concentration of the nutrient.

In addition to having direct pharmacological effects, IV nutrient therapy may be more effective than oral or IM treatment for correcting intracellular nutrient deficits. Some nutrients are present at much higher concentrations in the cells than in the serum. For example, the average magnesium concentration in myocardial cells is 10 times higher than the extracellular concentration. This ratio is maintained in healthy cells by an active-transport system that continually pumps magnesium ions into cells against the concentration gradient. In certain disease states, the capacity of membrane pumps to maintain normal concentration gradients may be compromised. In one study, the mean myocardial magnesium concentration was 65-percent lower in patients with cardiomyopathy than in healthy controls, (10) implying a reduction in the intracellular-to-extracellular ratio to less than 4-to-1. As magnesium plays a key role in mitochondrial energy production, intracellular magnesium deficiency may exacerbate heart failure and lead to a vicious cycle of further intracellular magnesium loss and more severe heart failure.

ELIGIBILITY:
Inclusion Criteria:

* N/A

Exclusion Criteria:

* N/A

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Urban or Rural
Sampling Method: Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2025-12-21 (Estimated); Primary Completion 2026-07-24 (Estimated); Study Completion 2026-09-17 (Estimated)

PRIMARY OUTCOMES:
Reduction in Symptoms related to Specific Illness or Disorder | 8-12 weeks, varying with each Intervention
  The percentage of patients who have lesser symptoms from their health issues and show measurable changes in heath, function, and quality of life that results from my care. I am creating a new supplement/vitamin brand that will reduce the symptoms of hypertension, anxiety, arthritis, fibromyalgia, nervousness and low energy levels among other conditions pertinent to herbal medicine and the patients involved in the study.

CONTACTS AND LOCATIONS:
Locations (1):
- Health for Life Holistic Wellness Center LLC, Dover, Delaware, United States

IPD SHARING:
Plan to Share IPD: Undecided